CLINICAL TRIAL: NCT06698406
Title: Transcultural Validation of the French Version of the " Patients' Endorsement of a Biopsychosocial Model of Chronic Pain " Scale
Status: Recruiting | Type: Observational
Sponsor: Benno Rehberg-Klug (Other)
Responsible Party: Sponsor-Investigator, Benno Rehberg-Klug, Clinical professor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: ABDC validation
Record Dates: First submitted 2024-11-18; First posted 2024-11-21 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Pain, Chronic
Keywords: pain, chronic; patient education; self efficacy; bio-psycho-social model
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We will validate the French version of the "Patients' Endorsement of a Biopsychosocial model of chronic pain (PEB) scale" by comparing it to the "pain self-efficacy" questionnaire

DETAILED DESCRIPTION:
The primary objective is to validate the French version of the PEB scale, called "Echelle d'Adhésion du modèle Bio-psycho-social par des patients avec Douleur Chronique ABDC".

The hypothesis is that the ABDC scale is a valid measurement tool to measure and operationalize beliefs about the biopsychosocial nature of pain in adults with chronic pain.

Consenting patients will receive paper copies of the study questionnaire including the questionnaires named in the secondary outcomes section, except those which are already included in the standard evaluation questionnaire of the pain consultation (BPI, GAD-7, PHQ-9). Patients will return the questionnaire either at a the same or a follow-up consultation, or send in the questionnaire by post in a prepaid envelope.

ELIGIBILITY:
Inclusion Criteria:

* - Patients with chronic pain (defined by ICD-11 as pain persisting or recurring longer than 3 months) having a chronic pain consultation at the HUG
* French-speaking and able to understand the study information
* ≥18 years of age

Exclusion Criteria:

* - Inability to understand the consent form and the questionnaire, e.g. due to lan-guage problems, psychological disorders, dementia, etc. of the participant
* Enrolment of the investigator, his/her family members, employees and other de-pendent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated by the ambulatory chronic pain clinic (consultation d'antalgie) of the HUG
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
incremental validity of the new ABDC scale | 1 day
  Incremental validity is the degree to which a new scale increases the ability to predict an outcome beyond existing parameters and scales. In our case pain self-efficacy, measured by the "pain self-efficacy questionnaire" [8], which exists in a validated French version [9], is the outcome to be predicted.
  Hierarchical regression analysis will have four models including in hierarchical order 8 explanatory variables: demographical variables (gender, age, level of education), depressive symptoms and anxiety, pain catastrophizing, pain acceptance, and finally the ABDC scale

SECONDARY OUTCOMES:
Reliability of the ABDC scale | 1 day
  Reliability will be evaluated as internal consistency, measured by Cronbach's alpha and corrected item-total-correlations.
Convergent validity | 1 day
  Convergent validity will be evaluated by the correlation between the ABDC scale sum score and the "Survey of Pain Attitudes SOPA" scale [10], a self-administered questionnaire with 57 statements evaluating 7 categories of beliefs and attitudes about pain.
Discriminant validity | 1 day
  correlations with the following scales which measure constructs which are important determinants of chronic pain severity, but independent of the endorsement of the biopsychosocial model by a patient: Brief Pain Inventory (BPI) The Brief Pain Inventory (BPI) [11] is a tool used to assess pain in patients. It was developed to measure both the intensity of pain and its impact on the patient's daily life. We will evaluate correlations with both the BPI-pain severity and the BPI-pain interference subscores.
  Generalized anxiety disorder questionnaire GAD-7 The GAD-7 [12] is a questionnaire used to assess generalized anxiety disorder. It consists of seven questions that evaluate different symptoms associated with anxiety, such as nervousness, restlessness, and difficulty controlling worry.
  Depressive symptoms: patient heath questionnaire PHQ-9 The PHQ-9 [13] is a screening tool for depression. It includes nine quest

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Genève, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No